CLINICAL TRIAL: NCT05874011
Title: Development of a Tool to Assess Receptive Prosody in the Aftermath of a Right Stroke: Use of the Inverse Correlation Paradigm
Brief Title: Prosody Assessment After Right Hemisphere Stroke
Acronym: ProsAVC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200144
Record Dates: First submitted 2023-05-05; First posted 2023-05-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Right Hemisphere Stroke
Keywords: Prosody; Reverse correlation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with right stroke consecutively recruited according to inclusion and non-inclusion criteria
  Interventions: Other: understanding of prosody
- Healthy volunteers: Healthy volunteers with no known history of stroke
  Interventions: Other: understanding of prosody

INTERVENTIONS:
Other: understanding of prosody — The inverse correlation test consists of having the same word heard twice, and asking which of the two sounds the most like a question. The exercise will be repeated several times, for a task that will take a total of about thirty minutes

SUMMARY:
Following a right stroke, more than half of the patients present a communication disorder. These disorders can notably concern prosody. Nevertheless, these remain relatively poorly assessed and characterized. Prosodic alterations in comprehension can result in a disruption of social cognition with potentially important consequences in terms of functional outcome and quality of life of patients. In clinical practice, the investigators do not have a tool that allows us to finely assess these disorders.

Studies in healthy subjects using a processing algorithm capable of arbitrarily manipulating the pitch dynamics of recorded voices have revealed that there are stable internal representations for prosody processing. Initial pilot results show that this method can be used in a clinical context and can indeed identify and accurately measure perceptual processing deficits in prosody following a right stroke. It is necessary to continue the study of this approach with a larger number of subjects in order to have normative data and validate the diagnostic properties of this approach.

DETAILED DESCRIPTION:
The aim of this project is to study impairments of speech prosodic perception using a novel data-driven psychoacoustic technique, reverse correlation.

The project will, first, conduct a prospective diagnostic study on N=150 stroke patients and controls, in order to evaluate the relevance of reverse-correlation data as a marker of prosodic impairments. Second, the project will use this novel patient data for theoretical investigations such as lesion-symptom mapping, in order to better understand how prosodic processing differs between patients and controls. Finally, the project will develop a novel mobile audio-health platform to facilitate the adoption of the reverse-correlation procedure in clinical practice and to collect remote patient data to assist medical decision-making.

The rationale of the reverse correlation technique is to uncover a listener's mental representation of certain prosodic patterns (e.g. the different intonation of "really?" vs "really!") by analyzing a large set of responses to random stimuli.

The expected results of the project are threefold: (1) the investigators will provide a new tool able to diagnose stroke-related prosody impairments beyond existing gold standards, (2) the investigators will provide a finer characterization of symptomatological profiles in these patients and (3) the investigators will provide a new prognosis metric, implemented in a mobile application, to quantify how well a patient reacts to speech therapy day after day.

The project will both further our understanding of aprosodia and provide new clinical tools to improve its diagnosis and rehabilitation. Beyond stroke, the project will also provide a case-study for the application of reverse-correlation to general speech therapy practice, benefiting patients across the whole spectrum of hearing impairments.

ELIGIBILITY:
-->Inclusion Criteria: Inclusion criteria for patients

Patient:

* with a right supratentorial stroke (1st clinical episode of deficit) confirmed on imaging and less than 1 year old at the time of inclusion
* right-handed
* male and female over 18 years of age
* french mother tongue
* affiliated or beneficiary of a social security plan
* free, informed and written consent signed
* Inclusion criteria for control subjects:

Subject:

* no known history of stroke
* right-handed
* over 18 years of age and matched with a case on age (plus or minus 10 years)
* french mother tongue
* affiliated or beneficiary of a social security plan
* free, informed and written consent signed

  -->Exclusion Criteria: Non-inclusion criteria for patients and controls subjects
* comprehension disorders: score less than 10/15 on the BDAE (Boston Diagnostic Aphasia Examination) command execution test
* known dementia
* illiteracy
* severe dysarthria
* psychiatric history requiring hospitalization in a specialized environment for more than two months
* history of brain injury
* major visual or auditory perceptual disorder (hearing loss greater than 40 dB HL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major patients with right supratentorial stroke and major control subjects with no known history of stroke will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-07-12 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Evolution of the inverse correlation task at the beginning and at the end of participation | 6 months
  The inverse correlation task that will be proposed in the study consists of presenting pairs of the word "really" with random variations in the height (F0) of the bounds of the six 71 ms segments of the word, asking them to distinguish within each pair which is the more interrogative.

SECONDARY OUTCOMES:
Assessment of musical perception | Inclusion, after 3 months and 6 months
  As the perception of prosody, whether linguistic or emotional, can be closely linked to musical perception, we will use the melodic part of the Montreal Amusia Assessment Battery (MBEA), considering the value of 65 as the pathological threshold, as established by the study by Peretz (Peretz, Champod, & Hyde, 2003).
Assessment of anxiety | Inclusion, after 3 months and 6 months
  Mood disorders following a stroke may influence the perception and production of prosody. In order to assess the presence of such disorders in the study subjects, we will use the HADS (Hospital and Anxiety Depression Scale) (Friedman, Samuelian, Lancrenon, Even, & Chiarelli, 2001; Zigmond & Snaith, 1983) which is a self-administered questionnaire composed of 14 questions on anxiety and depressive symptoms.
Assessment of depression | Inclusion, after 3 months and 6 months
  Mood disorders following a stroke may influence the perception and production of prosody. In order to assess the presence of such disorders in the study subjects, we will use the HADS (Hospital and Anxiety Depression Scale) (Friedman, Samuelian, Lancrenon, Even, & Chiarelli, 2001; Zigmond & Snaith, 1983) which is a self-administered questionnaire composed of 14 questions on anxiety and depressive symptoms.
Assessment of auditory attention | Inclusion, after 3 months and 6 months
  To determine whether or not attentional components are affected, we will use crossmodal integration and flexibility subtests from the Test of Attentional Performance (TAP, version 2.3.1, Zimmermann and Fimm, 2009).
Assessment of central auditory disorders | Inclusion, after 3 months and 6 months
  Difficulties in prosody perception may be due to central auditory disorders. Therefore, we will assess pitch, intensity and duration discrimination abilities using the AIRTAC2 software (Del Fabro & Desmons, 2014; Weill-Chounlamountry, Tessier, Soyez-Gayout, & Pradat-Diehl, 2010)
Assessment of hearing acuity | Inclusion, after 3 months and 6 months
  The hearing of the subjects will be measured by performing audiograms to ensure that there is no hearing loss.
Event-Related Potentials (EEG) | Inclusion, after 3 months and 6 months
  We will use an Electrical Geodesics device, consisting of a net of 256 electrodes wetted in a salt water solution and placed on the scalp; and a set of high impedance amplifiers connected to a Mac computer for digitising the signals. This is a method with excellent temporal resolution. Indeed, the entry into activity of a brain region is instantly accompanied by a tiny variation in electrical potential on the surface of the scalp, which the EEG amplifiers measure with extreme precision.
  Typically, we digitise EEG signals between 125 Hz and 500 Hz, which allows a temporal accuracy of 2 to 8 milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Marie VILLAIN, Ms., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.